CLINICAL TRIAL: NCT05936177
Title: Effects of 20 Minutes Osteoporosis Education on the Awareness of Osteoporosis in People Registered in Elderly Care Homes
Brief Title: Brief Osteoporosis Education to Increase Awareness in Middle Aged and Elderly.
Acronym: BOEIAMAE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selkin Yılmaz Muluk (Other Government)
Responsible Party: Sponsor-Investigator, Selkin Yılmaz Muluk, MD, Physical Therapy and Rehabilitation specialist, Antalya Training and Research Hospital
Organization: Antalya Training and Research Hospital (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 08.06.2023, no: 8/18
Record Dates: First submitted 2023-06-17; First posted 2023-07-07 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Osteoporosis
Keywords: osteoporosis; awareness; education; elderly
MeSH Terms: conditions — Osteoporosis | interventions — Patient Education as Topic

STUDY DESIGN:
Intervention Model Description: In this study, we plan to employ a statistical model as its primary framework for evaluation and analysis. The main focus of the study will center around the statistical modeling of data collected through pre and post-education questionnaires, as well as the demographic information of the participants and changes in their lifestyle habits. The study design will include cluster randomization, wherein two out of the four elderly homes in our municipality will be randomly selected using a simple random sampling technique (via coin toss) to be part of the study. Participants attending to these selected houses will be recruited as volunteers through short message service (SMS) invitations. This approach will enable us to examine and analyze the impact of the education intervention on participants' knowledge levels, as well as their potential shifts in lifestyle choices.
Masking Description: The study does not involve masking for participants, investigator and assessors as the primary objective is to assess the impact of pre and post-education interventions on awareness scores, which are objective measures not subject to potential bias from knowledge of the intervention status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Education Group (Other): The Education Group arm will involve participants who receive the osteoporosis education intervention, which includes a concise educational session delivered by a physiatrist, covering various topics related to osteoporosis. Participants in this arm will have the opportunity to enhance their knowledge and awareness of osteoporosis through the provided educational materials and interactive discussions.
  Interventions: Other: Patient education

INTERVENTIONS:
Other: Patient education — The intervention in this osteoporosis education research will consist of a concise and informative educational session delivered by a physiatrist, utilizing slides prepared based on information from reputable sources such as the International Osteoporosis Foundation website and the World Health Organization (WHO) health education booklet. The session will cover various topics including the definition of osteoporosis, its causes, risks, complications, dietary options, and specific exercise recommendations, with a focus on raising awareness and promoting informed decision-making regarding prevention and treatment options.
  Other Names: Not present

SUMMARY:
Osteoporosis is a growing global concern, particularly as the population of middle-aged and elderly individuals continues to rise within communities. This demographic, being more susceptible to chronic diseases, poses a burden on healthcare systems. The objective of this study is to explore methods of educating middle-aged and elderly individuals about osteoporosis, aiming to raise awareness of the disease and promote informed decision-making regarding prevention and treatment options

DETAILED DESCRIPTION:
This research will involve visiting all four Elderly Houses in Muratpasa, Antalya. After obtaining informed consent, participants will be asked to provide demographic information, including age, sex, and education levels, as well as relevant medical history, such as family history of osteoporosis. Additionally, participants will complete a validated questionnaire called the Osteoporosis Knowledge Assessment Tool (OKAT).

Those who express interest in further education will be enrolled in an osteoporosis education program, which will be scheduled accordingly. The education program will utilize slides prepared based on information from the International Osteoporosis Foundation website (http://www.osteoporosis.foundation) and the WHO health education booklet. Delivered by a physiatrist, the education session will be concise, lasting approximately 20 minutes, and will cover various topics, including the definition of osteoporosis, its causes, risks, complications, dietary options, and specific exercise recommendations.

Following the education session, participants will once again complete the OKAT questionnaire to assess any changes in knowledge. They will also have the opportunity to have their questions addressed. One month later, participants will be contacted by phone for a follow-up interview, during which changes in their dietary habits, sun exposure, exercise routines, and other relevant factors will be discussed. Lastly, participants will complete the OKAT questionnaire for the third time.

These measures will help evaluate the effectiveness of the osteoporosis education intervention and provide insights into any potential changes in participants' knowledge and behavior over time.

ELIGIBILITY:
Inclusion Criteria:

1. Middle-aged and elderly individuals (e.g., 50 years and above).
2. Ability to understand and communicate in the language of the study materials (Turkish).
3. Willingness to participate in the study and provide informed consent.
4. Residency in the community where the Elderly Houses are located (Muratpasa, Antalya).
5. Availability to attend the education session and complete follow-up assessments.

Exclusion Criteria:

1. Severe cognitive impairments or mental health conditions that may hinder comprehension or participation.
2. Pre-existing knowledge or educational background in osteoporosis, particularly through careers in health systems, that may bias the results.
3. Participation in any other osteoporosis education programs within a specified period before the study.
4. Inability to complete the questionnaire independently or engage in follow-up communication.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2023-06-08 (Actual); Primary Completion 2023-09-29 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
Change in participants' knowledge about osteoporosis. | Pre-education assessment (baseline) and immediate post-education assessment (short-term)
  Change in participants' knowledge about osteoporosis before and after the education. This can be assessed using the Osteoporosis Knowledge Assessment Tool. Each correct answer receives 1 point, and incorrect or unknown answers receive 0 points, resulting in scores ranging from 0 to 20, based on this 20-question questionnaire. High scores mean a better awareness.

SECONDARY OUTCOMES:
Changes in participants' exercise habits. | Pre-education assessment (baseline) and one month follow-up assessment (medium-term).
  Does the education cause increase in participants' exercise routines?
Changes in participants' dietary habits. | Pre-education assessment (baseline) and one month follow-up assessment (medium-term).
  Does the education cause increase in participants' calcium intake?
Changes in participants' sun exposure habits. | Pre-education assessment (baseline) and one month follow-up assessment (medium-term).
  Does the education cause an increase in participants' duration of sun exposure?

CONTACTS AND LOCATIONS:
Overall Officials: Selkin Yılmaz, Principal Investigator — Antalya Ataturk Devlet Hastanesi
Locations (1):
- Elderly Homes (Fener, Soğuksu, Konuksever, Ciftekuyular Yaslı Evleri), Antalya, Muratpasa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The IPD sharing plan for this osteoporosis education study prioritizes participant confidentiality and privacy. Therefore, the individual participant data will not be openly or publicly shared due to ethical considerations and the sensitive nature of the data. However, we support transparency and scientific collaboration.
  Upon request, deidentified aggregate data or summary statistics may be shared with qualified researchers for collaborative research, meta-analyses, or further exploration of study outcomes. Data sharing will comply with data protection regulations and guidelines.
  Requests for data access will be evaluated case-by-case by the principal investigator and research team, considering scientific validity, participant privacy protection, and ethical principles. Data access may require appropriate data sharing agreements and compliance with institutional and ethical review board policies.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: October 2023-October 2024
Access Criteria: Access to the individual participant data (IPD) will be granted to qualified researchers or institutions engaged in scientific research or analysis related to osteoporosis education.
  Researchers must comply with ethical guidelines and data protection regulations.
  Researchers must sign a data use agreement and submit a research proposal outlining their study objectives and methodology.
  Access to the IPD will be subject to review and approval by an access committee or data sharing board.
  No data access fee will be charged.

REFERENCES:
- [Background] Gai QY, Lv H, Li YP, Fu QM, Li P. Education intervention for older adults with osteoporosis: a systematic review. Osteoporos Int. 2020 Apr;31(4):625-635. doi: 10.1007/s00198-019-05166-5. Epub 2019 Dec 11. PMID 31828364
- [Background] Jensen AL, Lomborg K, Wind G, Langdahl BL. Effectiveness and characteristics of multifaceted osteoporosis group education--a systematic review. Osteoporos Int. 2014 Apr;25(4):1209-24. doi: 10.1007/s00198-013-2573-5. Epub 2013 Nov 23. PMID 24270886
- [Background] Rubaek M, Hitz MF, Holmberg T, Schonwandt BMT, Andersen S. Effectiveness of patient education for patients with osteoporosis: a systematic review. Osteoporos Int. 2022 May;33(5):959-977. doi: 10.1007/s00198-021-06226-5. Epub 2021 Nov 12. PMID 34773131
- [Background] Kalkim A, Daghan S. Theory-based Osteoporosis Prevention Education and Counseling Program for Women: A Randomized Controlled Trial. Asian Nurs Res (Korean Soc Nurs Sci). 2017 Jun;11(2):119-127. doi: 10.1016/j.anr.2017.05.010. Epub 2017 Jun 28. PMID 28688497
- [Background] Etemadifar MR, Nourian SM, Fereidan-Esfahani M, Shemshaki H, Nourbakhsh M, Zarezadeh A. Relationship of knowledge about osteoporosis with education level and life habits. World J Orthop. 2013 Jul 18;4(3):139-43. doi: 10.5312/wjo.v4.i3.139. Print 2013 Jul 18. PMID 23878783
- [Background] Sayed-Hassan R, Bashour H, Koudsi A. Osteoporosis knowledge and attitudes: a cross-sectional study among female nursing school students in Damascus. Arch Osteoporos. 2013;8:149. doi: 10.1007/s11657-013-0149-9. Epub 2013 Sep 3. PMID 23999904
- See also: The information presented in the PowerPoint slides has been derived from the 'International Osteoporosis Foundation' website. — https://www.osteoporosis.foundation/patients
- Available data/document: Health education concepts and strategies: World Health Organization — https://apps.who.int/iris/bitstream/handle/10665/119953/EMRPUB_2012_EN_1362.pdf?sequence=1&isAllowed=y

DOCUMENTS (1):
  • Informed Consent Form (2023-06-08): https://cdn.clinicaltrials.gov/large-docs/77/NCT05936177/ICF_000.pdf